CLINICAL TRIAL: NCT06214494
Title: Effects of Blood Flow Restricted High Intensity Treadmill Training on Independently Ambulating Chronic Ischemic CVA Survivors: A Pilot Study
Brief Title: Blood Flow Restricted High-Intensity Treadmill Training on Independently Ambulating Chronic Ischemic CVA Survivors
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: MedStar National Rehabilitation Network (Other)
Responsible Party: Principal Investigator, Jane Alkhazov, Principal Investigator, MedStar National Rehabilitation Network
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BFR-HITT
Record Dates: First submitted 2023-12-29; First posted 2024-01-19 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-03

CONDITIONS: Stroke, Ischemic; Ambulation Disorder, Neurologic; Chronic Stroke
Keywords: Blood Flow Restriction Training; BFR; BFRt; High Intensity Treadmill Training
MeSH Terms: conditions — Ischemic Stroke; Gait Disorders, Neurologic

STUDY DESIGN:
Intervention Model Description: A Randomized Case Control Cohort Study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Interventional Cohort (Experimental): Blood Flow Restricted High Intensity Treadmill Training at 70% limb occlusion 2x weekly for 16 Sessions totaling a minimum of 75 minutes weekly.
  Interventions: Other: Blood Flow Restricted High Intensity Treadmill Training
- Control Cohort (Active Comparator): High-Intensity Treadmill Training 2x weekly for 16 Sessions totaling a minimum of 75minutes weekly.
  Interventions: Other: HITT

INTERVENTIONS:
Other: Blood Flow Restricted High Intensity Treadmill Training — Blood Flow Restricted High Intensity Treadmill Training at 70% limb occlusion (on hemiparetic limb only) 2x weekly for 16 Sessions totaling minimum of 75 minutes weekly.
  Other Names: BFR-HITT
  Arms: Interventional Cohort
Other: HITT — High Intensity Treadmill Training 2x weekly for 16 Sessions totaling minimum of 75minutes weekly.
  Arms: Control Cohort

SUMMARY:
Individuals surviving Chronic Ischemic Stroke have lingering walking deficits long after their infarct. The main goal of this study is to compare two high intensity treadmill walking programs to see which improves walking more. The main question we aim to answer is: How does blood flow restricted high-intensity treadmill training impact walking function? Participants will be randomly separated into two groups. One group will perform the high intensity treadmill training with blood flow restriction on their Stroke affected leg, while the second group performs high intensity treadmill training only. Every week participants will be asked to walk on the treadmill for a total of 75 minutes during 2x 1-hour sessions. On visit 1, participants will undergo strength, balance, and walking testing. They will then be treated 2x weekly for 4 weeks (visit 2-9) and be re-tested to track progress on visit 10. Participants will again be treated 2x weekly for 4 more weeks (visit 11-18) and be tested to see the end results on visit 19. Researchers will then compare both groups to see if blood flow restriction training changes walking function, strength, and balance.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years or older with history of single ischemic stroke >6months.
* Ambulate without physical assistance over 10M with or without mobility aides and bracing in 180 seconds or less.

Exclusion Criteria:

* Concurrent physical or occupational therapy.
* Vulnerable populations such as adults unable to consent, individuals who are not yet adults (infants, children, teenagers), pregnant women, prisoners will be excluded.
* Resting BP >160/100mmHg even with medication.
* People who have taken analgesics, dopamine, antipyretics, and any other drugs that can affect the function of the autonomic nervous system in the last 2 weeks and likely to be treated with such drugs during the course of the study.
* Individuals who score 9 (greater than normal or minimal impairment) or more on the Short Blessed Cognitive Assessment (6 item) will be unable to give informed consent.
* Any medical condition (including heart failure, unstable angina, aortic stenosis, arrhythmias, hypertrophic cardiomyopathy, depression of ST-segment, previous or active deep vein thrombosis (DVT) in the hemiparetic lower extremity, pulmonary embolism (PE), bypass surgery within last 3 months.) that, in the opinion of the investigator, might jeopardize the participants' safety.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
6 Minute Walk Test | Baseline, Week 4 (up to one week), Week 8( up to one week)
  The 6-minute walk test (6MWT) assesses distance walked over 6 minutes as a sub-maximal test of aerobic capacity/endurance.

SECONDARY OUTCOMES:
10 Meter Walk Test | Baseline, Week 4 (up to one week), Week 8( up to one week)
  The 10MWT assesses walking speed in meters per second over a short duration.
5 Time Sit to Stand | Baseline, Week 4 (up to one week), Week 8( up to one week)
  The Five Times Sit to Stand Test measures one aspect of transfer skill. The test provides a method to quantify functional lower extremity strength and/or identify movement strategies a patient uses to complete transitional movements.
Functional Gait Assessment | Baseline, Week 4 (up to one week), Week 8( up to one week)
  The FGA is used to assess postural stability during walking and assesses an individual's ability to perform multiple motor tasks while walking. The tool is a modification of the 8-item Dynamic Gait Index, developed to improve reliability and reduce ceiling effect. Each item is scored on an ordinal scale from 0 to 3, with 0 = severe impairment, 1 = moderate impairment, 2 = mild impairment, 3 = normal ambulation. The highest score = 30 indicating no impairment in postural stability during walking.
BERG Balance Scale | Baseline, Week 4 (up to one week), Week 8( up to one week)
  The Berg Balance Scale (BBS) is a 14-item objective measure that assesses static balance and fall risk in adults. Item-level scores range from 0-4 and are determined by ability to perform the assessed activity Item scores are then summed with lower scores indicating higher fall risk. The maximum score = 56.
Activities Balance Confidence Scale-16 | Baseline, Week 4 (up to one week), Week 8( up to one week)
  The ABC Scale is a self-report measure of balance confidence in performing various activities without losing balance or experiencing a sense of unsteadiness. Items are rated on a rating scale that ranges from 0 - 100. Score of zero represents no confidence, a score of 100 represents complete confidence.
  Overall score is calculated by adding item scores and then dividing by the total number of items.

OTHER OUTCOMES:
Lower Extremity Limb Circumference | Baseline, Week 4 (up to one week), Week 8( up to one week)
  Limb circumference (cm) of hemiparetic lower extremity and unaffected lower extremity will be taken to determine if limb hypertrophy has occurred.
1 Repetition Maximum Strength Testing (Leg press) | Baseline, Week 4 (up to one week), Week 8( up to one week)
  1 Repetition Maximum Strength Testing (Leg press) is a measure of overall hemiparetic gross push strength and is measured as the greatest force (in lbs) a patient can push with hemiparetic lower extremity one time.
1 Repetition Maximum Strength Testing (Knee Extension) | Baseline, Week 4 (up to one week), Week 8( up to one week)
  1 Repetition Maximum Strength Testing (Knee Extension) is a measure of isolated hemiparetic quadriceps strength and is measured as the greatest force (in lbs) a patient can extend their hemiparetic quadriceps one time.

CONTACTS AND LOCATIONS:
Locations (1):
- MedStar National Rehabilitation Hospital, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No